CLINICAL TRIAL: NCT00332839
Title: Multi-center, Open-label, Prospective, Randomized, Parallel Group Study Investigating a CNI-free Regimen With Enteric-coated Mycophenolate Sodium and Everolimus in Comparison to Standard Therapy With Enteric-coated Mycophenolate Sodium and Ciclosporin Microemulsion in Stable Renal Transplant Patients
Brief Title: Comparison of CNI-based Regimen Versus CNI-free Regimen in Kidney Transplant Recipients.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The trial was terminated early due to slow enrollment. It was determined that the planned sample size of 300 could not be achieved.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRAD001ADE02; 2005-001013-18
Record Dates: First submitted 2006-05-31; First posted 2006-06-02 (Estimated); Results first posted 2014-08-28 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Renal Transplantation
Keywords: enteric-coated mycophenolate sodium, everolimus, CNI-free regimen
MeSH Terms: interventions — Everolimus; Cyclosporine; Tacrolimus; Mycophenolic Acid; Adrenal Cortex Hormones

ARMS (2):
- Calcineurin Inhibitor (CNI) group (Active Comparator): Participants received Cyclosporine A (CsA) plus Enteric Coated Mycophenolate Sodium (EC-MPS) plus corticosteroids, or Tacrolimus A (CsA) plus Enteric Coated Mycophenolate Sodium (EC-MPS) plus corticosteroids.
  Interventions: Drug: Cyclosporin A (CsA); Drug: Tacrolimus; Drug: Enteric Coated - Mycophenolate Sodium (EC-MPS); Drug: Corticosteroids
- Certican group (Experimental): Participants were switched in a step-wise fashion from the CNI based regimen to Everolimus (RAD001).
  Interventions: Drug: Everolimus; Drug: Enteric Coated - Mycophenolate Sodium (EC-MPS); Drug: Corticosteroids

INTERVENTIONS:
Drug: Everolimus — Participants, switching from the CsA based treatment, initially received everolimus 1.5 mg/day and then from day 7, 3 mg/day, and then from day 14, the dose was based on the participants' blood level (6-10 ng/ml). Participants, switching from the tacrolimus based treatment, initially received 3 mg/day and then from day 14, the dose was based on the participants' blood level (6-10 ng/ml).
  Other Names: RAD001, Certican
  Arms: Certican group
Drug: Cyclosporin A (CsA) — The dose was based on the participants' blood level of C0h (80-150 ng/ml).
  Other Names: Sandimmun Optoral
  Arms: Calcineurin Inhibitor (CNI) group
Drug: Tacrolimus — The dose was based on the participants' blood level of C0h (5-10 ng/ml).
  Other Names: Prograf
  Arms: Calcineurin Inhibitor (CNI) group
Drug: Enteric Coated - Mycophenolate Sodium (EC-MPS) — The dose was ≥ 720 mg/day.
  Other Names: Myfortic
Drug: Corticosteroids — Corticosteroids were given according to local standard and/or the Investigators' discretion.

SUMMARY:
Calcineurin inhibitors (CNI), a potent immunosuppressive drug used in kidney transplant recipients to prevent graft rejection, may cause renal impairment. The aim of this study is to assess whether a CNI-free regimen with enteric-coated mycophenolate sodium and everolimus is as safe and well tolerated as a standard regimen consisting of enteric-coated mycophenolate sodium and cyclosporine microemulsion without a compromise in therapeutic efficacy while resulting in an improved renal function.

ELIGIBILITY:
Inclusion Criteria:

Males or females, aged > 18 years, Maintenance renal transplant recipients at least 6 months post-transplantation, Patients with a serum creatinine < 2,5 mg/dL stable for at least three month (according to the investigator), Females capable of becoming pregnant had to have a negative serum pregnancy test within seven days prior to or at baseline, and were required to practice an approved method of birth control for the duration of the study and for a period of six weeks following discontinuation of study medication, even where there had been a history of infertility, Patients receiving Myfortic® (Myfortic dose . 720 mg/d) and Sandimmun® Optoral with or without corticosteroids as part of their immunosuppressive regimen for at least 1 month before baseline;

Exclusion Criteria:

More than one previous renal transplantation, Multi-organ recipients (e.g., kidney and pancreas) or previous transplant with any other organ, different from kidney, Patient with proteinuria > 1000 mg/day at baseline, Hypersensitivity to Certican®, Sandimmun® Optoral, Prograf®, mycophenolic acid, or other components of the formulation, Patients who had received an investigational drug within four weeks prior to baseline, Severe rejection (≥ Banff II acute rejection), recurrent acute rejection, or steroid resistant rejection within six months of enrollment, Thrombocytopenia (platelets < 100,000/mm³), with an absolute neutrophil count of < 1,500/mm³ or leukopenia (leukocytes < 4,000/mm³), or hemoglobin < 8 g/dL, Abnormal physical or laboratory findings of clinical significance within two weeks of study inclusion which at the investigator's discretion would interfere with the objectives of the study, Symptoms of significant somatic or mental illness. Inability to cooperate or communicate with the investigator, or patients who were unlikely to comply with the study requirements, or who were unable to give informed consent, History of malignancy during the last five years, except squamous or basal cell carcinoma of the skin, Patients who were HIV positive, or hepatitis C, or hepatitis B surface antigen positiveEvidence of severe liver disease (including abnormal liver enzyme profile, i.e. aspartate transaminase (AST), alanine aminotransferase (ALT) or total bilirubin > 3 times upper limit of normal (ULN), Females of childbearing potential who were planning to become pregnant, who were pregnant or lactating and/or who were unwilling to use effective means of contraception, Presence of a clinically significant infection requiring continued therapy, severe diarrhea, active peptic ulcer disease or uncontrolled diabetes mellitus that in the opinion of the investigator would interfere with the appropriate conduct of the study, Evidence of drug or alcohol abuse

Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2005-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis, Study Director — Novartis
Locations (10):
- Germany (10):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Heilbronn
  - Novartis Investigative Site, Kaiserslautern
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Münster

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Renal transplant recipients at least 6 months post transplantation were randomized to the CNI group or Certican group. Post 12 months, participants entered a follow-up phase for an additional 48 months. Thirty-three participants in the CNI group and 34 participants in the Certican group had a month 60 follow-up status.
Period: Core (Months 0 - 12)
Arm/Group | Calcineurin Inhibitor (CNI) Group | Certican Group
Started | 47 | 46
Safety Set | 47 | 46
Completed | 37 | 28
Not Completed | 10 | 18
Not completed — Administrative problems | 1 | 1
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Protocol deviation | 1 | 1
Not completed — Adverse Event | 5 | 15
Period: Follow-up (Months 12 - 60)
Arm/Group | Calcineurin Inhibitor (CNI) Group | Certican Group
Started | 33 (Follow-up included core participants (completed or discontinued) who wished to be followed.) | 34 (Follow-up included core participants (completed or discontinued) who wished to be followed.)
Completed | 29 | 31
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Death | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Calcineurin Inhibitor (CNI) Group | Certican Group | Total
Number analyzed (Participants) | 47 | 46 | 93
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.8 (11.1) | 51.0 (10.3) | 50.4 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 17 | 29
  Male | 35 | 29 | 64

OUTCOME MEASURES:

1. Primary Outcome: Renal Function
Description: The analysis for this outcome measure was not perfomed because the analyses could not be powered for efficacy due to low recruitment.
Time Frame: 12 months
Arm/Group | Calcineurin Inhibitor (CNI) Group | Certican Group
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Biopsy Proven Acute Rejection, Graft Loss, and Death
Description: as for outcome 1
Time Frame: 12 months
Arm/Group | Calcineurin Inhibitor (CNI) Group | Certican Group
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Occurrence of Treatment Failures
Description: as for outcome 1
Time Frame: 12 months
Arm/Group | Calcineurin Inhibitor (CNI) Group | Certican Group
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Evolution of Renal Function
Description: as for outcome 1
Time Frame: Baseline, 12 months
Arm/Group | Calcineurin Inhibitor (CNI) Group | Certican Group
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants Who Experienced Adverse Events and Death
Description: Participants were monitored for adverse events, serious adverse events and deaths thorughout the prospective and follow-up phases of the study.
Time Frame: 12 months
Population: The safety set, which included all randomized participants, comprised the analysis population.
Measure: Number; unit: Participants
Arm/Group | Calcineurin Inhibitor (CNI) Group | Certican Group
Number analyzed (Participants) | 47 | 46
Participants
  Adverse events (serious and non-serious) | 44 | 44
  Serious adverse events | 11 | 12
  Deaths | 1 | 1

6. Secondary Outcome: Changes in Cardiovascular Risk
Description: as for outcome 1
Time Frame: Baseline, 12 months
Arm/Group | Calcineurin Inhibitor (CNI) Group | Certican Group
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Changes in Proteinuria
Description: as for outcome 1
Time Frame: Baseline, 12 months
Arm/Group | Calcineurin Inhibitor (CNI) Group | Certican Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Calcineurin Inhibitor (CNI) Group | Certican Group
Serious Adverse Events (participants affected / at risk) | 11/47 | 12/46
Other Adverse Events (participants affected / at risk) | 31/47 | 41/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Calcineurin Inhibitor (CNI) Group (N=47) | Certican Group (N=46)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Multi-organ failure (General disorders) | 0 | 1
Nodule (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Abscess (Infections and infestations) | 1 | 0
Cystitis klebsiella (Infections and infestations) | 0 | 1
Cytomegalovirus colitis (Infections and infestations) | 1 | 1
Cytomegalovirus gastroenteritis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 0 | 1
Proteus infection (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 3
Wound infection (Infections and infestations) | 0 | 1
Wound infection staphylococcal (Infections and infestations) | 0 | 1
Graft dysfunction (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Transplant failure (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 2 | 0
Blood human chorionic gonadotropin increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1
Migraine without aura (Nervous system disorders) | 1 | 0
Albuminuria (Renal and urinary disorders) | 0 | 1
Calculus bladder (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Testicular disorder (Reproductive system and breast disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Calcineurin Inhibitor (CNI) Group (N=47) | Certican Group (N=46)
Anaemia (Blood and lymphatic system disorders) | 3 | 8
Leukopenia (Blood and lymphatic system disorders) | 2 | 6
Abdominal pain (Gastrointestinal disorders) | 5 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 12
Diarrhoea (Gastrointestinal disorders) | 10 | 7
Oedema peripheral (General disorders) | 3 | 11
Nasopharyngitis (Infections and infestations) | 11 | 11
Urinary tract infection (Infections and infestations) | 1 | 5
Blood creatine phosphokinase increased (Investigations) | 1 | 6
Blood creatinine increased (Investigations) | 8 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 5
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 6
Proteinuria (Renal and urinary disorders) | 3 | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 8
Acne (Skin and subcutaneous tissue disorders) | 1 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 5

LIMITATIONS AND CAVEATS:
Adverse Events data were not collected during the Follow-up period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.